CLINICAL TRIAL: NCT04606706
Title: Development and Effectiveness of A Mobile Health-Based Education Intervention on Maternal, Infant and Young Child Nutrition to Prevent Stunting in Kelantan
Brief Title: A mHealth Based Education Intervention on Maternal, Infant and Young Child Nutrition to Prevent Stunting in Kelantan
Acronym: stunting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Norshafawati Binti Abd. Azimi, Principal investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 311/PPSK/4117626
Record Dates: First submitted 2020-09-14; First posted 2020-10-28 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Mobile Health; Healthy
Keywords: Mobile health; Education intervention; Maternal; Infant; Young child; Nutrition; Stunting
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal, lactating mother & young child (Intervention) (Experimental): mHealth education intervention for 6 months
  Interventions: Other: Mobile health nutrition education intervention
- Maternal, lactating mother & young child (Control) (No Intervention): Conventional health education

INTERVENTIONS:
Other: Mobile health nutrition education intervention — Nutrition education will be given through mobile phone
  Arms: Maternal, lactating mother & young child (Intervention)

SUMMARY:
This research aimed to develop health module related to nutrition through mobile phone and to access it effectiveness among mother, infant and children (0-2 years old) to prevent stunting in Kelantan, Malaysia. Besides, to evaluate the effectiveness of intervention in reducing stress among pregnant and lactating women. The mobile health (mHealth) messaging interventions will be delivered via a mobile app known as WhatsApp and by a phone call. There will be a total of 50 messages for 6 months of intervention in which 2 messages will be delivered per week (every Tuesday & Thursday). The understanding of information will be evaluated 2 times per month by a phone call. The type of messages that will be used are text messages, voice messages, video/graphic messages, and voice calls. The assessment using a brief questionnaire and anthropometry measurement will be conducted during first and at the end of the intervention. The effectiveness and perceptions as well as experiences of mobile health intervention will also be assessed.

DETAILED DESCRIPTION:
A) Research Objectives

1. General Objective

   To evaluate the effectiveness of mobile health intervention program and to explore the perceptions and experiences of mobile health intervention among mothers to prevent stunting among infant and young children in Kelantan, Malaysia
2. Specific Objectives

Phase 1 - Development of a mobile health education package to prevent stunting among maternal, infant and young children

1. To develop the mobile health education package for pregnant women, lactating mothers and mothers of young children in preventing stunting among children

   Phase 2 - Evaluation of the effectiveness of mobile health intervention program to prevent stunting
2. To compare the changes in anthropometric measurement and dietary intake after 6 months of intervention among pregnant women, lactating mothers, infants and children in Kelantan
3. To compare the changes in knowledge, attitude and practice of breastfeeding after 6 months of intervention among lactating mothers

   Phase 3 - Qualitative study
4. To explore the perceptions and experiences of mobile health intervention among lactating mothers and their husband

B) Study Location

This study will be conducted in selected 6 districts in Kelantan, Malaysia which are Jeli, Gua Musang, Kuala Krai, Tanah Merah, Pasir Mas and Kota Bharu

C) Sample Size

Sample size for each study group (pregnant women, lactating mothers and children) were calculated by using G-power software.

Total sample size for each group = 150 subjects After including 15% of dropout compensation, the final total sample size calculated for each group of this study = 172 subjects Thus, the total sample size for each arm (intervention and control groups) for each group of study = 86 subjects

For face-to-face interview, subjects will be recruited until saturation is achieved. An estimated 20-30 subjects will be recruited in this study (Mason, 2010). The face-to-face interview will be audio recorded.

D) Population and Sampling Method

This study will involve antenatal mothers with husband, lactating mothers with infant and husband, and children's with mother that will be selected by using multistage sampling method

E) Research Tools

1. Questionnaire

   1. Socio-demographic and socio-economic questionnaire
   2. Belief toward feeding practice questionnaire
   3. Validated food security questionnaire i. 10 items Radimer/Cornell hunger scale
2. Nutrient intake questionnaire i. 3-days 24-hour diet recall
3. Validated mental health questionnaire i. Depression, anxiety and stress scale
4. Validated knowledge, attitude and practice on breastfeeding and infant and young child feeding questionnaire
5. Programme satisfaction questionnaire

F) Anthropometric measurement instrument:

1. Baby weighing scale
2. Adult weighing scale
3. Height measuring scale
4. Measuring tape
5. Body composition analyzer

G) mHealth Intervention Package

All the messages will be created in Malay language based on the books, booklets, topics and modules that have been developed by World Health Organization (WHO) 2012 and UNICEF 2012, and also have widely and officially used by Ministry of Health Malaysia to educate their patients. Basically, the source of messages that will be created and use are from:

1. Knowledge on breastfeeding (based on 13 breastfeeding topics for antenatal and postnatal)
2. Knowledge on infant and young child feeding (10 key messages for complementary feeding by WHO 2012 & key messages booklets for Infant and Young Child Feeding (IYCF) practices from UNICEF, 2012 in simplified form)
3. Knowledge on bottle handling and bottle feeding
4. Knowledge on formula milk preparation
5. Knowledge on hand washing
6. Information on healthy nutrition intake

H) mHealth Mode of Intervention

Intervention will be conducted by using a mobile phone. Thus, a "call centre" for this mobile health intervention program will be set up in Universiti Sains Malaysia (USM) Health Campus. All the information about breastfeeding, infant and young child feeding, bottle handling and bottle feeding, formula milk preparation, hand washing and nutrition intake will be disseminate through a mobile apps known as WhatsApp and by a phone call. There will be a total of 50 messages for 6 months of intervention which are 2 messages per week (every Tuesday & Thursday). The understanding of information will be evaluate 2 times per month by a phone call. The type of messages that will be used are:

1. Text messages
2. Voice messages
3. Video/graphic messages
4. Voice calls

A child growth chart (height) also will be give to respondents with infants and children.

I) Data Collection Procedure

Data collection will be conducted at selected districts and health clinics after obtaining approval from USM Research Ethics Committee and Medical Research and Ethics Committee, Ministry of Health Malaysia. This intervention study will be conducted over 6 months. All of the subjects who meet the inclusion and exclusion criteria will be recruited from the health clinics and will be referred to the call center of this study by a trained nutritionist. The purpose of the study and the randomization process will be explained to the subjects by a nutritionist during subjects recruitment.

All subjects (wife and husband only) will sign the informed consent form and parents permission form (for infant and children). The baseline and after 6 months of intervention data will be collected by a researcher and research assisstants of this study while a face-to-face interview will be collected by a researcher. Thus, this research will involve several procedures for mother, children and husband/father.

Mother:

Each mother will involve in anthropometric measurement (including body weight, height/length, body composition) and have to answer the questionnaire during the first and at the end of the intervention sessions.The questionnaire consist of sosio-demography, sosio-economy, medical history, belief toward food intake, food security, nutrient intake, mental health, knowledge, attitude and practice of breastfeeding and infant nutrition and children, and satisfaction of the programme. The estimate time taken to complete the questionnaire is 30 minutes.

For each mother selected in group 2, additional health related information will be provided periodically through mobile phone for 6 months. Health education information also will be given conventionally at health clinic. Whereas mother in group 1 will receive health education information conventionally at health clinic for 6 months. The subjects will be randomly assigned. The selected subject will also be interviewed at the end of the study.

Children:

All children involved will undergo anthropometric measurements (body weight, length, body composition) during the first and at the end of intervention.

Husband/Father:

For husband/father whom their spouse are selected in group 2, additional health related information will be provided periodically through mobile phone for 6 months. Health education information also will be given conventionally at health clinic. Whereas husband/father whom their spouse are selected in group 1 will receive health education information conventionally at health clinic for 6 months. A few husband/father whom their spouse selected to be interviewed also will be interviewed at the end of intervention.

Each interview will take about 40 to 60 minutes to complete.

Group 1 - Control group; Group 2 - Intervention group

ELIGIBILITY:
Inclusion Criteria:

Pregnant women + husband

1. Malaysian
2. Pregnant women age 18-35 years during the study
3. Height (<155 cm)
4. or B40 (household income below Ringgit Malaysia (RM) 2194 in Kelantan)
5. or history of stunted child
6. or History Gestional Diabetes Mellitus (GDM), anemia, pre-eclampsia
7. In second trimester of pregnancy (13-16 weeks)
8. Attend the same selected health clinics for the regular medical check-up
9. Own a smart phone

Lactation mother + infant + husband

1. Malaysian
2. Lactation mother age 18-35 years during the study
3. Mother height (<155 cm)
4. or B40 (household income below RM 2194 in Kelantan)
5. or history of stunted child
6. New postnatal cases reported to the clinic after delivery
7. Attend the selected health clinics for the regular medical check-up
8. Own a smart phone

Children + mother + father

1. Malaysian
2. Children age 6-18 months
3. B40 (household income below RM2194 in Kelantan)
4. or stunted siblings
5. Full terms' babies (deliver after 37 weeks gestation)
6. Attend the selected health clinics for the regular medical check-up
7. Own a smart phone

Exclusion Criteria:

Pregnant women + husband

1) Multiple pregnancies

Lactation mother + infant + husband

1. Babies who have congenital problems/ birth defects
2. Stillbirth or foetal death after deliver

Children + mother + father

1. Children who have congenital problems/ birth defects
2. Single parent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 516 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight after 6 months of intervention among mother, infant and children | 6 months
  Body weight in kg
Changes in body mass index after 6 months of intervention among mother, infant and children | 6 months
  Body mass index in kg/m^2
Changes in body composition after 6 months of intervention among mother, infant and children | 6 months
  Body composition in %
Changes in dietary intake after 6 months of intervention among mother, infant and children | 6 months
  24-hour diet recall (3-days) in kcal
Assessment of food security level after 6 months of intervention among mother, infant and children | 6 months
  Food security in score (All items are negative answer = secure; If one or more item have positive answer = insecure)
Assessment of mental stress after 6 months of intervention among mother, infant and children | 6 months
  Mental stress in score (Depression if score >9; anxiety if score > 7; stress if score > 14)
Assessment of socioeconomic status (SES) after 6 months of intervention among mother, infant and children | 6 months
  Socioeconomic status (SES) in Ringgit Malaysia unit

SECONDARY OUTCOMES:
Changes in knowledge, attitude and practice of breastfeeding after 6 months of intervention among lactating mothers | 6 months
  Total score of knowledge in percentage (A higher percentage means good knowledge), Higher score of attitude means positive attitude

OTHER OUTCOMES:
Perceptions on mobile health intervention among lactating mothers and their husband | after 6 months
  Perceptions on mobile health (qualitative-based)
|Experiences on mobile health intervention among lactating mothers and their husband | after 6 months
  Experiences on mobile health (qualitative-based)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No